CLINICAL TRIAL: NCT07090642
Title: Effectiveness of Digital Escape Room Game-Based Disaster Midwifery Training: MERCI Model
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, YASEMİN AYDIN KARTAL, Prof. Dr., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: SBU-AYDINKARTAL-AKER
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-07

CONDITIONS: Digital Escape Room; Game-Based Learning
Keywords: Disaster midwifery; digital escape room; clinical decision making; game-based learning; self-efficacy

STUDY DESIGN:
Intervention Model Description: Randomized controlled double-blind experimental study
Who Masked: Participant, Investigator
Masking Description: The research process will be conducted with a double-blind design; both participants and data collectors will be unaware of group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (Experimental): Simultaneously with the module training, the four-part escape room game "M.E.R.C.I." will be applied to the intervention group.
  Interventions: Other: Digital escape room game
- Control group (No Intervention): In addition to standard theoretical training, case-based learning techniques will be applied to students in the control group.

INTERVENTIONS:
Other: Digital escape room game — Concurrent with the module training, the intervention group will be given the four-part escape room game "M.E.R.C.I." The game's sections will be developed in parallel with the weekly topics of the disaster midwifery module training.
  Arms: İntervention group

SUMMARY:
Midwives play important societal roles during the post-crisis transition and recovery phase. Specific guidelines regarding the roles and responsibilities of midwives, who constitute a significant majority among healthcare professionals, in disaster management need to be developed, and the concept of disaster midwifery needs to be developed. Providing midwife candidates with disaster awareness throughout their undergraduate education will also positively impact individuals' self-efficacy. In recent years, educational plans for emergency obstetric care and management have evolved from traditional theoretical and clinical training to game-based learning, gamification, and training using mannequins and simulators. It is suggested that using different learning strategies in the training of healthcare professionals in emergency obstetric situations will improve the quality of care and reduce maternal mortality rates. Natural disasters such as disasters can cause serious obstetric emergencies requiring immediate intervention and management. Supporting the professional training of midwives, who play important roles and responsibilities in disaster management, with diverse teaching strategies is crucial for enhancing their individual competencies.

This study is based on a game-based learning approach through an interactive, educational digital escape room game developed on the Genially platform. Therefore, this study was designed to investigate the effects of a digital escape room game-based disaster midwifery training on midwifery students' knowledge, self-efficacy in disaster response, and confidence and anxiety levels in clinical decision-making. This experimental study, designed with a randomized pretest, posttest, and follow-up design and a control group, will be conducted with third- and fourth-year midwifery students in the Department of Midwifery at the Health Sciences University (SBU), Hamidiye Faculty of Health Sciences (HSBF), during the spring semester of the 2025-2026 academic year. The sample size was determined using Koca and Arkan's study. Based on a Cohen's d = 1.35 effect size and a power level of 95%, a total of 80 participants were planned, with 40 students in each group. Participants included in the study will be administered the "Informed Consent Form," "Introductory Information Form," "Disaster Midwifery Information Form," "Disaster Intervention Self-Efficacy Scale," "Self-Confidence and Anxiety Scale in Clinical Decision Making," and "Game Experience Scale." Discussions and conclusions of the study will be written based on the findings.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study.
* Having internet access.
* Having a smartphone.
* Having successfully completed a course on normal birth and postpartum.
* Being an active third-year student in the Midwifery Department of Hamidiye Faculty of Health Sciences, University of Health Sciences.
* Being an active fourth-year student in the Midwifery Department of Hamidiye Faculty of Health Sciences, University of Health Sciences.

Exclusion Criteria:

* Being a 4th-year inactive student in the Midwifery Department of Hamidiye Faculty of Health Sciences, University of Health Sciences.
* Being a 3rd-year inactive student in the Midwifery Department of Hamidiye Faculty of Health Sciences, University of Health Sciences.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | 10 minitus
  This form, created by researchers based on literature, includes questions about the participants' age, high school graduation, their self-sufficiency against disasters, etc.
Disaster Midwifery Information Form | 20 minitus
  This form was developed by researchers based on literature and based on the content of the disaster midwifery module used as a theoretical training module. The final version will be finalized based on expert opinion. Twenty multiple-choice questions were prepared, deemed appropriate for the research purpose and educational content. The form's performance will be evaluated out of 100 points. For this purpose, students' total success scores are calculated as five times the number of correct answers. Students will be evaluated by assigning "5" points for each correct answer and "0" points for each incorrect answer. The highest possible score for students on the information form is "100," and the lowest is "0."
Disaster Response Self-Efficacy Scale | 20 minitus
  Developed by Hong-Yan Li and his colleagues in 2017 and its Turkish validity safety studies were conducted by Koca et al. in 2018, the Disaster Response Self-Efficacy Scale consists of 19 items and 3 sub-dimensions and the responses were taken using a 5-point Likert scale. A high score on the scale indicates a high level of disaster response self-efficacy. The scale has three sub-factors. Sub-factors are: "On-Site Rescue Competence (Items 1 - 11)", "Disaster Psychological Nurse Competence (Items 12 - 15)" and "The nature of the role undertaken in disaster and adaptation adequacy (Items 16 - 19)". The Cronbach alpha coefficient for the entire scale is 0.96. The Cronbach alpha values obtained for the sub-dimensions are; On-site rescue competence was determined as 0.93, psychological nurse competence in disaster was determined as 0.93, and the quality of the role undertaken in the disaster and adaptation competence was determined as 0.93 (Bennur et al., 2020).
Nursing Anxiety and Self-Confidence with Clinical Decision Making (NASC-CDM) Scale | 20 minitus
  The scale, which provides separate scores for self-confidence and anxiety, is a 6-point Likert-type scale consisting of 27 questions. The scale has three subscales for both the self-confidence and anxiety sections: "using sources to obtain information and listening fully," "using available information to identify the problem," and "knowing and taking action." Increasing scores in the self-confidence and subscales indicate increasing students' self-confidence in clinical decision-making. Low scores in the anxiety section and its subscales indicate low anxiety levels in clinical decision-making. The lowest possible score for the self-confidence and anxiety sections is 27, and the highest is 162. The total Cronbach alpha coefficient of the self-confidence section of the scale is 0.97, and the total Cronbach alpha coefficient of the anxiety section is 0.96 (Bektaş et al., 2017).

SECONDARY OUTCOMES:
Disaster Midwifery Information Form | 20 minitus
  This form was developed by researchers based on literature and based on the content of the disaster midwifery module used as a theoretical training module. The final version will be finalized based on expert opinion. Twenty multiple-choice questions were prepared, deemed appropriate for the research purpose and educational content. The form's performance will be evaluated out of 100 points. For this purpose, students' total success scores are calculated as five times the number of correct answers. Students will be evaluated by assigning "5" points for each correct answer and "0" points for each incorrect answer. The highest possible score for students on the information form is "100," and the lowest is "0."
Disaster Response Self-Efficacy Scale | 20 minitus
  Disaster Response Self-Efficacy Scale: Developed by Hong-Yan Li and his colleagues in 2017 and its Turkish validity safety studies were conducted by Koca et al. in 2018, the Disaster Response Self-Efficacy Scale consists of 19 items and 3 sub-dimensions and the responses were taken using a 5-point Likert scale. A high score on the scale indicates a high level of disaster response self-efficacy. The scale has three sub-factors. Sub-factors are: "On-Site Rescue Competence (Items 1 - 11)", "Disaster Psychological Nurse Competence (Items 12 - 15)" and "The nature of the role undertaken in disaster and adaptation adequacy (Items 16 - 19)". The Cronbach alpha coefficient for the entire scale is 0.96. The Cronbach alpha values obtained for the sub-dimensions are; On-site rescue competence was determined as 0.93, psychological nurse competence in disaster was determined as 0.93, and the quality of the role undertaken in the disaster and adaptation competence was determined as 0.93.
Nursing Anxiety and Self-Confidence with Clinical Decision Making Scale | 20 minitus
  Description: The scale, which provides separate scores for self-confidence and anxiety, is a 6-point Likert-type scale consisting of 27 questions. The scale has three subscales for both the self-confidence and anxiety sections: "using sources to obtain information and listening fully," "using available information to identify the problem," and "knowing and taking action." Increasing scores in the self-confidence and subscales indicate increasing students' self-confidence in clinical decision-making. Low scores in the anxiety section and its subscales indicate low anxiety levels in clinical decision-making. The lowest possible score for the self-confidence and anxiety sections is 27, and the highest is 162. The total Cronbach alpha coefficient of the self-confidence section of the scale is 0.97, and the total Cronbach alpha coefficient of the anxiety section is 0.96 (Bektaş et al., 2017).
Gaming Experience Scale (Only the intervention group) | 20 minitus
  The validity and reliability study of the scale was conducted by Dönmez et al. in 2024. This scale, adapted for nursing students, aims to assess individuals' experiences while playing digital games. The 27-item scale consists of five subscales: enjoyment (items 1-6), immersion (7-12), creative thinking and emotional activation (13-17, 19-20), absence of negative effects (18, 21-23), and mastery (24-27). Evaluation is made using a 5-point Likert-type scale (1 = Never, 5 = Always), and items 18, 21, 22, and 23 are reverse-scored. The structure obtained in the exploratory factor analysis supports validity; the scale's overall Cronbach's alpha internal consistency coefficient is 0.93. Alpha values for the subscales range from 0.78 to 0.93. High scores indicate that the individual has a more enjoyable, participatory and satisfying gaming experience (Dönmez et al., 2024).

OTHER OUTCOMES:
Disaster Midwifery Information Form | 20 minitus
  This form was developed by researchers based on literature and based on the content of the disaster midwifery module used as a theoretical training module. The final version will be finalized based on expert opinion. Twenty multiple-choice questions were prepared, deemed appropriate for the research purpose and educational content. The form's performance will be evaluated out of 100 points. For this purpose, students' total success scores are calculated as five times the number of correct answers. Students will be evaluated by assigning "5" points for each correct answer and "0" points for each incorrect answer. The highest possible score for students on the information form is "100," and the lowest is "0."

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No